CLINICAL TRIAL: NCT01905475
Title: CXCR4 AnTagonism for Cell Mobilisation and Healing in Acute Myocardial Infarction (CATCH-AMI). A Phase IIa, Double-Blind, Placebo-Controlled, Randomised, Multi-centre Study of POL6326, a CXCR4 Antagonist, in Patients With Large Reperfused ST Elevation Myocardial Infarction
Brief Title: CXCR4 Antagonism for Cell Mobilisation and Healing in Acute Myocardial Infarction (CATCH-AMI)
Acronym: CATCH-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POL6326-POL-006
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Large Reperfused ST-Elevation Myocardial Infarction
Keywords: STEMI; AMI; repair
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — balixafortide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- POL6326 (Experimental): POL6326 intravenous infusion
  Interventions: Drug: POL6326
- Placebo (Placebo Comparator): Placebo intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: POL6326
  Arms: POL6326
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of POL6326 (CXCR4 antagonist) as a stem cell mobilizing agent, on cardiac function and infarct size and on safety and tolerability, in patients with reperfused ST-Elevation Myocardial Infarction (STEMI).

DETAILED DESCRIPTION:
After acute myocardial infarction and successful stent implantation patients will undergo a baseline MRI (magnetic resonance imaging) for eligibility for the study. Patients will receive POL6326 or placebo in the first week after STEMI. The primary and secondary endpoints will also be determined in a follow-up visit after 12 months. An interim analysis will be performed after 50% of the patients have completed the 4 months MRI assessment and may result in an adjustment of study size. A number of pre-specified subgroups will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms suggestive of an acute MI with ST-segment elevation or new left bundle-branch block and a rise or fall in cardiac necrosis markers.
2. Patients must be scheduled to undergo coronary angiography for the purposes of primary PCI (percutaneous coronary intervention) culminating in successful stent implantation.
3. Age between 18 and 80 years. Male and WOCBP (women of child bearing potential) willing to use highly effective methods of contraception from the time of first dose until 3 months after the last dose of the drug.
4. Markedly reduced LVEF at baseline cardiac MRI.
5. No previous occurrence of Myocardial Infarction.
6. Estimated glomerular filtration rate (eGFR) equal or higher than 40 mL/minute prior to MRI.
7. Signed Informed Consent.

Exclusion Criteria:

1. Evidence of multi-vessel coronary artery disease likely to require repeat PCI or coronary artery bypass grafting within 4 months.
2. Pulmonary oedema or cardiogenic shock requiring intubation or mechanical support at the time of the planned baseline MRI.
3. Fitted with a non-MRI-compatible cardiac pacemaker or implantable cardioverter defibrillator, or expected to require such a device within 4 months after randomisation.
4. Terminal illness or malignant disease.
5. Advanced hepatic disease.
6. Diagnosis of severe obesity which precludes MRI assessments.
7. Claustrophobia.
8. Acute systemic infection or fever.
9. Anemia (where hemoglobin levels are <10 g/dL), thrombocytopenia (platelet count <100000/μL) or coagulopathy.
10. History of multiple drug allergies or with a known allergy to the drug class of CXCR4 antagonists.
11. Pregnancy or females of childbearing potential who are not using double contraception
12. Known history of human immunodeficiency virus (HIV) infection, chronic hepatitis B or hepatitis C infection or significant active chronic inflammatory disease that requires immunosuppressive medication or regular systemic corticosteroids.
13. Patients who have participated in any investigational drug or device trial within 30 days prior to signing informed consent.
14. Patients who are unwilling or unable to abide by the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in LVEF (left ventricular ejection fraction) as determined by MRI | 4 months
  Difference in LVEF from baseline (after STEMI and stent procedure, before infusion of drug or placebo) and after 4 months

SECONDARY OUTCOMES:
Additional measures of cardiovascular function | 4 months
  Using MRI the following parameters will also be determined: infarct size, LV volumes, regional LV function. Plasma BNP (brain natriuretic peptide) will also be determined.
Mobilization of stem and progenitor cells | 2 days
  Time dependent measurement of stem and progenitor cells during and after infusion of POL6326
Pharmacokinetic outcome | 2 days
  Measurement of plasma concentrations of POL6326 at predose and several time points after infusion.
Safety of POL6326 by intravenous infusion | 12 months
  Safety as measured by incidence, type and severity of adverse events (Major Adverse Cardiovascular Events (MACE), Arrhythmia)

CONTACTS AND LOCATIONS:
Overall Officials: Kai C. Wollert, MD, Principal Investigator — Hannover Medical School
Locations (17):
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna
- Germany (4):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Charité - Campus Benjamin, Berlin
  - Charité - Campus Virchow, Berlin
  - Hannover Medical School, Hanover
- Hungary (6):
  - Semmelweis University, Budapest
  - Magyar Honvédség Egészségügyi Központ, Kardiológiai osztály, Budapest
  - DEOEC, Kardiológiai Intézet, Debrecen
  - Kaposi Mór Teaching Hospital, Kaposvár
  - Pécs University, Pécs
  - Zala Megyei Kórház,Kardiológia, Zalaegerszeg
- Hospital John Paul II, Krakow, Poland
- United Kingdom (4):
  - Edinburgh Heart Centre Royal Infirmary, Edinburgh
  - West of Scotland Regional Heart & Lung Center, Golden Jubilee National Hospital, Glasgow
  - University Hospitals of Leicester NHS Trust Glenfield Hospital, Leicester
  - King's College Hospital, London